CLINICAL TRIAL: NCT06825728
Title: Metoprolol in Patients With Heart Failure With Reduced Ejection Fraction and Chronic Obstructive Pulmonary Disease
Brief Title: Metoprolol in Patients With HFrEF and COPD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202412231; 2022YFC2010004 (Other Grant/Funding Number: National key research and development plan)
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Heart Failure with Reduced Ejection Fraction; Chronic Obstructive Pulmonary Disease; Metoprolol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group received the maximum tolerable dose of Metoprolol.
  Interventions: Drug: Different doses of Metoprolol.
- Control Group (Active Comparator): The control group received 23.75mg/d of Metoprolol.
  Interventions: Drug: Different doses of Metoprolol.

INTERVENTIONS:
Drug: Different doses of Metoprolol. — The control group received 23.75mg/d of metoprolol, and the experimental group received the maximum tolerable dose of metoprolol.

SUMMARY:
The goal of the clinical trial was to see if Metoprolol was effective in treating patients with heart failure and chronic obstructive pulmonary disease. It will also learn about the safety of Metoprolol. The main questions it aims to answer are:

Did Metoprolol reduce the frequency of all-cause deaths and re-hospitalizations in subjects? What medical problems do participants experience after taking Metoprolol? The researchers will compare different doses of Metoprolol to see the best dose for Metoprolol.

Participants will:

Take Metoprolol 23.75mg/ day or the maximum tolerable dose of Metoprolol daily for 24 months.

Regular outpatient follow-up visits to the research center. Their symptoms and Metoprolol dosage were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. A definite diagnosis of HFrEF (LVEF≤40%), NYHA II to IV , and the disease is due to ischemic heart disease or dilated cardiomyopathy;
2. A definite diagnosis of COPD with moderate or higher airflow limitation (FEV1/FVC < 0.7 and FEV1 < 80% of the expected value);
3. Age ≥18 years old;
4. Informed consent has been obtained and signed.

Exclusion Criteria:

1. the dose of Metoprolol before enrollment was more than 23.75mg/d;
2. Resting heart rate < 50 beats/min;
3. Second or third degree atrioventricular block;
4. Atrial fibrillation;
5. Sick sinus syndrome;
6. Systolic blood pressure < 90mmHg;
7. Acute attack of bronchial asthma;
8. Liver insufficiency (serum transaminase > 3 times the normal value);
9. Renal insufficiency (eGFR < 30ml/min/1.73m2, or serum creatinine > 2.5mg/dL[> 221μmol/L]);
10. Patients with serious physical diseases, such as cancer;
11. Patients who have a history of allergy to the investigational drug or its ingredients;
12. Participating in other clinical investigators;
13. During the study period, Patients cannot live in the selected center for a long time, which is not conducive to the follow-up;
14. Patients with disability, mobility disability, intellectual disability and other factors that may prevent normal participation in the study and follow-up, and their frailty was assessed by the FRAIL frailty screening scale; Intellectual mental status was assessed by the Mini-Mental State Examination (MMSE).
15. Poor adherence or other reasons considered by the researchers to be unsuitable for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Composite endpoints (all-cause death and rehospitalization) | From enrollment to the end of treatment at 24 months.
  Rehospitalization included readmission for heart failure and/or COPD.

SECONDARY OUTCOMES:
All-cause death | From enrollment to the end of treatment at 24 months.
Cardiovascular death | From enrollment to the end of treatment at 24 months.
Rehospitalization for heart failure | From enrollment to the end of treatment at 24 months.
Re-hospitalization for COPD | From enrollment to the end of treatment at 24 months.